CLINICAL TRIAL: NCT00318721
Title: Efficacy, Acceptability and Cost-effectiveness of Long Lasting Insecticide Nets (LLIN) in the Prevention of Kala Azar
Acronym: KALANET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); University Hospital, Geneva (Other); Rajendra Memorial Research Institute of Medical Sciences (Other); Institute of Medical Sciences of the Banaras Hindu University, India (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Prof Marleen Boelaert, Institute of Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CT-2005-015374
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-06

CONDITIONS: Visceral Leishmaniasis; Kala Azar
Keywords: Leishmania donovani; cluster-randomised control trial; Long Lasting Impregnated Nets; Bednets; Sandflies
MeSH Terms: conditions — Leishmaniasis, Visceral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: Long Lasting Impregnated Nets (LLIN)
- control (No Intervention)
  Interventions: Device: Long Lasting Impregnated Nets (LLIN)

INTERVENTIONS:
Device: Long Lasting Impregnated Nets (LLIN) — Distribution of LLIN in selected clusters

SUMMARY:
A cluster-randomized vector control trial in Bihar, India, and neighboring Nepal, will test the efficacy of long-lasting impregnated bednets (LLINs, Permanets) for reducing visceral leishmaniasis incidence. The intervention unit is the village (400-1000 people). The study is designed to detect a 50% reduction in Leishmania donovani incidence in intervention compared to control clusters over 2 years. 24 clusters (selected as high incidence during previous years) will be randomly allocated to intervention or control. Following health education, and with informed consent, all households in intervention villages will receive free Permanets (from September 2006). Net usage will be monitored and new nets provided if required. Control villages will not be given untreated nets, as - although commonly used in this region - their effectiveness against sandflies has not been proven. Pre-intervention infection status of villagers (>2 yrs) will be evaluated serologically from finger-prick blood (and past/current disease status noted). Incident infections will be recorded by 3-monthly active search for clinical cases, and by annual serological diagnoses to detect subclinical infections. All villagers (>2yrs) will be leishmanin skin tested at the end of the trial for further subclinical infection detection, and sera from a sub-sample will be tested for antibodies to sandfly saliva antigens (a measure of sandfly exposure). All clinical cases will be given free treatment. Free Permanets will be provided to control villages after the trial. Complementary studies involve entomological surveillance by light traps in a sample of houses and social/economic questionnaire surveys. The entomological surveys will test whether community-wide use of LLINs provides any mass effect, which could protect those in the community who fail to use LLIN for any reason.

ELIGIBILITY:
Inclusion criteria (Clusters):

1. at least have seen 1 case per year in each of the last 3 years
2. An average of at least 1% Incidence rate over the period of past 3 years.

Exclusion criteria (Clusters):

1. Minimum 500 people
2. Maximum 2000 people
3. Distance between clusters 2000 meters (distance between borders)
4. Houses in tola/ward not sprayed (DDT, other) in 2006
5. Accessibility

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
L. donovani infection | yearly

SECONDARY OUTCOMES:
Kala Azar cases | quarterly

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Boelaert, Dr, Principal Investigator — Prince Leopold Institute of Tropical Medicine in Antwerp (ITM), Belgium; Clive Davies, Dr., Principal Investigator — London School of Hygiene and Tropical Medicine; Jean Claude Dujardin, Dr, Principal Investigator — Prince Leopold Institute of Tropical Medicine in Antwerp (ITM), Belgium; Suman Rijal, Dr., Principal Investigator — B.P. Koirala Institute of Heath Sciences, Nepal; Shyam Sundar, Dr, Principal Investigator — Institute of Medical Sciences of the Banaras Hindu University, India; Francois Chappuis, Dr., Principal Investigator — University Hospital, Geneva; Beena Varghese, Dr, Principal Investigator — Centre for Health and Population Research (ICDDR,B), Dhaka, Bangladesh; Marc Coosemans, Dr, Principal Investigator — Prince Leopold Institute of Tropical Medicine in Antwerp (ITM), Belgium.; Veerle Vanlerberghe, Dr., Principal Investigator — Prince Leopold Institute of Tropical Medicine in Antwerp (ITM), Belgium.; Diwarkar Dinesh, Dr, Principal Investigator — Rajendra Memorial Research Institute of Medical Sciences
Locations (2):
- Kala Azar Medical Research Center, Muzaffarpur, Bihar, India
- B P Koirala Institute of Health Sciences, Dharān, Nepal

REFERENCES:
- [Derived] Picado A, Das ML, Kumar V, Kesari S, Dinesh DS, Roy L, Rijal S, Das P, Rowland M, Sundar S, Coosemans M, Boelaert M, Davies CR. Effect of village-wide use of long-lasting insecticidal nets on visceral Leishmaniasis vectors in India and Nepal: a cluster randomized trial. PLoS Negl Trop Dis. 2010 Jan 26;4(1):e587. doi: 10.1371/journal.pntd.0000587. PMID 20126269